CLINICAL TRIAL: NCT06096129
Title: Cholangioscopy With Spyglass DS Using Percutaneous Transhepatic Cholangiography Access: a Retrospective Cohort Study
Brief Title: Cholangioscopy With Spyglass DS Using Percutaneous Transhepatic Cholangiography Access
Acronym: Spy PTC
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Trygve Ulvund Solstad, MD (Medical Doctor), Rigshospitalet, Denmark
Other Study IDs: R-21069569
Record Dates: First submitted 2023-10-05; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Biliary Stricture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spy PTC: People who had Spy PTC performed
  Interventions: Procedure: Spy PTC

INTERVENTIONS:
Procedure: Spy PTC — Percutaneous transhepatic cholangioscopy with SpyGlass DS system

SUMMARY:
Conventional peroral methods to visualize biliary strictures are not feasible in some patients with altered anatomy or biliary obstruction, and percutaneous transhepatic cholangioscopy can be used as an alternative procedure. This study aimed to retrospectively review the use of percutaneous transhepatic cholangiography using the SpyGlass DS technology (S-PTCS) during a 5-year period at a Danish tertiary referral center.

DETAILED DESCRIPTION:
Biliary strictures are caused by various disorders ranging from inflammatory strictures induced by primary sclerosing cholangitis (PSC) to strictures caused by cholangiocarcinoma. Identifying the etiology of these strictures is often difficult, but important, as treatment is dependent on the underlying cause1-3. To properly treat and diagnose biliary strictures, visualization of the target area is needed, and biopsies must be taken3,4. Conventional methods have poor accuracy in distinguishing between benign and malignant etiologies, and diagnosing these patients presents a challenge1,4,5.

Endoscopic retrograde pancreatography (ERCP) is the standard procedure for the treatment of biliary strictures1 and can be further supplemented with magnetic resonance cholangiopancreatography to increase diagnostic accuracy. However, ERCP is limited by its low diagnostic sensitivity6. Furthermore, some difficult strictures require direct visualization of the lesions with targeted biopsies. In such cases, peroral cholangioscopy (POCS) provides an alternative when traditional ERCP is not feasible. POCS can directly visualize target lesions, obtain targeted biopsies, and is shown to be safe and useful when diagnosing indeterminate biliary strictures1. However, some patients have previously undergone upper gastrointestinal surgery, which can alter both duodenal and biliary anatomy. Moreover, strictures caused by PSC may be multifocal and/or positioned over the biliary confluence, which can make visualization difficult2. Conventional ERCP and POCS are not feasible in these patients, and another approach is required7,8.

Percutaneous transhepatic cholangioscopy (PTCS) is an alternative, attractive procedure owing to a shorter and more straightforward route to all parts of the biliary tree. Studies have shown that PTCS is safe, effective, and feasible for the visualization of indeterminate biliary strictures and in cases with altered biliary anatomy7,9-12. In addition, the studies demonstrated high diagnostic accuracy of PTCS and reported a satisfactory rate of technical success7,9-12.

Despite these preliminary studies, literature concerning the feasibility of PTCS using SpyGlass DS technology (S-PTCS) remains sparse. This study aimed to evaluate the use, specifically the visual and histological success, and the specificity, sensitivity, and complication rate of S-PTCS during a 5-year period at a Danish tertiary referral center for upper gastrointestinal and hepato-pancreato-biliary surgery and transplantation.

ELIGIBILITY:
Inclusion Criteria:

* People above the 18 who underwent Spy PTC in this 5 year period

Exclusion Criteria:

* People under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See above
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Success in terms of finding diagnosis | baseline, 1 month after the procedure, follow up 4 or more years later
  Success rate of Spy PTC finding diagnosis later verified through histopathology/scans

SECONDARY OUTCOMES:
Safety in terms of complications | during the procedure, up to one month after procedure
  Number of participants with complications after procedure requiring intervention in general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, MD, Ph.D, Study Director — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The plan is to publish the study in a international medical journal.
Supporting Information: CSR
Time Frame: The information will be published in a medical journal sometime during the next two years.
Access Criteria: Will be entered when accepted in a journal.